CLINICAL TRIAL: NCT04342689
Title: The Role of Resistant Starch in COVID-19 Infection
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to low enrollment.
Sponsor: Yale University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Sherry Mansour, Instructor of Medicine, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000027887
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Results first posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
Keywords: COVID-19; Resistant Starch; Inflammation
MeSH Terms: conditions — COVID-19; Inflammation | interventions — Resistant Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects will receive a dietary supplement containing resistant starch and be instructed to take 2 tablespoons (~20 grams) twice daily for 14 days. Initially subjects will take 2 tablespoons once daily for the first three days prior to increasing to 2 tablespoons twice daily.
  Interventions: Drug: Dietary Supplement containing resistant starch
- Control (Placebo Comparator): Subjects will receive a placebo starch, consisting of non resistant starch and be instructed to take 2 tablespoons (~ 20 grams) twice daily for 14 days. Initially subjects will take 2 tablespoons once daily for the first three days.
  Interventions: Dietary Supplement: Placebo Starch

INTERVENTIONS:
Drug: Dietary Supplement containing resistant starch — Two tablespoons (~ 20 grams) to be taken twice daily for 14 days (start with 2 tablespoons once daily for three days, followed by twice daily on days 4 through 14)
  Other Names: Resistant Starch
  Arms: Intervention
Dietary Supplement: Placebo Starch — Two tablespoons (~ 20 grams) to be taken twice daily for 14 days (start with 2 tablespoons once daily for three days, followed by twice daily on days 4 through 14)
  Other Names: Non Resistant Starch
  Arms: Control

SUMMARY:
This study is a multicenter randomized trial to evaluate the efficacy of administering a dietary supplement containing resistant starch to non-hospitalized COVID-19 positive subjects, The intervention will begin as soon as possible after subjects test positive for COVID-19 and continue for 14 days. Investigators hypothesize that short-term administration of a dietary supplement containing resistant starch has the potential to reduce rates of hospitalization and improve time to clinical recovery and symptoms in non-hospitalized COVID-19 positive patients.

DETAILED DESCRIPTION:
The COVID-19 pandemic has caused a substantial strain on the healthcare system, with at least 14% of infected patients requiring hospitalization. Identifying ways to ameliorate the progression and severity of the COVID-19 infection and preventing hospitalization is critical. Patients suffering from COVID-19 have been shown to have a significant inflammatory response resembling that of cytokine release syndrome, and it is this inflammatory phase that is thought to drive fatality.

To this end, a multi-center randomized clinical trial to determine the efficacy of resistant starch in reducing the need for hospitalization for COVID-19 positive patients will be studied. This study will enroll 1500 non-hospitalized COVID-19 positive individuals who are being monitored in the outpatient setting. Patients will be randomized to either a dietary supplement containing resistant starch or a placebo for 14 days. Our primary outcome is the rate of hospitalization for COVID-19 related complications. Secondary outcomes will look at time to recovery and symptom severity scores.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years of age
* COVID-positive status
* Being monitored in an outpatient setting at one of our study sites:
* Yale New Haven Hospital (YNHH)
* University of Michigan
* University of Minnesota

Exclusion Criteria:

* inflammatory bowel disease
* history of gastric bypass surgery
* active Clostridium difficile infection
* active participation in another COVID-19 interventional trial
* any physical or psychological condition that, in the opinion of the investigator, would pose unacceptable risk to the patient or raise concern that the patient would not comply with the protocol procedures.
* Reported allergy to starch
* Difficulty swallowing in order to prevent any aspiration risk
* Currently taking any IL-6 inhibitors such as Tocilizumab for any disease condition

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Mansour, MD, MS, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data underlying results for publication are planned to be made available after publication.
Supporting Information: Study Protocol, SAP
Time Frame: After publication, indefinitely

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Supplement: Subjects will receive a placebo starch, consisting of non resistant starch and be instructed to take 2 tablespoons (~ 20 grams) twice daily for 14 days. Initially subjects will take 2 tablespoons once daily for the first three days.
  Placebo Starch: Two tablespoons (~ 20 grams) to be taken twice daily for 14 days (start with 2 tablespoons once daily for three days, followed by twice daily on days 4 through 14)
- Resistant Starch Supplement: Subjects will receive a dietary supplement containing resistant starch and be instructed to take 2 tablespoons (~20 grams) twice daily for 14 days. Initially subjects will take 2 tablespoons once daily for the first three days prior to increasing to 2 tablespoons twice daily.
  Dietary Supplement containing resistant starch: Two tablespoons (~ 20 grams) to be taken twice daily for 14 days (start with 2 tablespoons once daily for three days, followed by twice daily on days 4 through 14)
Period: Overall Study
Arm/Group | Placebo Supplement | Resistant Starch Supplement
Started | 113 | 113
Completed | 71 | 68
Not Completed | 42 | 45
Not completed — Withdrawal by Subject | 32 | 33
Not completed — Lost to Follow-up | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Supplement | Resistant Starch Supplement | Total
Number analyzed (Participants) | 113 | 113 | 226
Age, Continuous [Median (Full Range); unit: years] | 45 [19 to 77] | 45 [19 to 79] | 45 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 70 | 135
  Male | 48 | 43 | 91
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 92 | 94 | 186
  White | 15 | 13 | 28
  Unknown | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 113 | 113 | 226

OUTCOME MEASURES:

1. Primary Outcome: Count of Participant Hospitalization for a COVID-19 Related Complication (Phase 3)
Description: Hospitalization for a COVID-19 related admission during the first month of follow up. Death prior to hospitalization thought to be secondary to COVID-19 will also be defined as an event.
Time Frame: One month from the start of treatment
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 113 | 113
Participants | 2 | 2
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.99, Chi-squared

2. Secondary Outcome: Time to Clinical Recovery (TTCR) (Phase 2)
Description: Time to clinical recovery will be defined by a return to normal body temperature (97-99 degrees F) as reported by the patient, and resolution of major presenting symptoms (myalgia, cough, shortness of breath, and GI symptoms) maintained for 72 hours. Patients will be called every 2 days for the first 14 days of the study, and then once weekly for the following 14 days to assess symptoms via a pre-specified questionnaire. Patients will be followed from the start of treatment to the end of follow-up at 4 months.
Time Frame: One month from the start of treatment, up to 4 months
Population: Intention to treat
Measure: Median (Full Range); unit: days
Arm/Group | Resistant Starch Supplement | Placebo Supplement
Number analyzed (Participants) | 113 | 113
days | 12 [0 to 42] | 8 [0 to 42]
Statistical Analysis 1: Comparison: Resistant Starch Supplement vs Placebo Supplement; Test type: Superiority; p = 0.52, t-test, 2 sided

3. Secondary Outcome: Peak Symptom Severity Score (Phase 2)
Description: This score will be evaluated using a subjective self-reporting questionnaire around 8 symptoms, which include: shortness of breath at rest or exertion, fatigue, myalgia/muscle aces, fever, cough, headache, GI symptoms, inability to taste or smell. Subjects will rate each of their symptoms on an ordinal scale as follows: absent (0), mild (1), moderate (2), or severe (3). These symptom ratings will be added to define the symptom severity score with a possible score range of 0-24 points. Subjects will be called every 2 days for the first 14 days of the study, and then once weekly for the following 14 days to assess symptoms via this pre-specified questionnaire. Patients will be followed from the start of treatment to the end of follow-up at 4 months. "Peak" was added to the outcome title (to correctly identify the measure) when results were entered.
Time Frame: One month from the start of treatment, up to 4 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Resistant Starch Supplement | Placebo Supplement
Number analyzed (Participants) | 113 | 113
score on a scale | 6 [0 to 16] | 5 [0 to 17]
Statistical Analysis 1: Comparison: Resistant Starch Supplement vs Placebo Supplement; Test type: Superiority; p = 0.24, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 1 month after completion of treatment course
Arm/Group | Placebo Supplement | Resistant Starch Supplement
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/113
Other Adverse Events (participants affected / at risk) | 24/113 | 35/113
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Supplement (N=113) | Resistant Starch Supplement (N=113)
Gas (Gastrointestinal disorders) | 24 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT04342689/Prot_SAP_000.pdf